CLINICAL TRIAL: NCT05942235
Title: Effect of mıcro learnıng Based Wound healıng Course on clınıcal reasonıng skılls of nursıng Students
Brief Title: The Use of Microlearning in Nursing Education
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Yasemin GÜNER, lecturer, Karadeniz Technical University
Other Study IDs: 123456
Record Dates: First submitted 2022-12-20; First posted 2023-07-12 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Nursing Education; Wound Healing; Educational Problems
Keywords: Nursing Education; Wound Healing; Active Learning
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control grup 1: Among the students enrolled in the surgical diseases nursing course in the fall semester, 42 students will be selected using the "research randomizer" program. Then, students will be asked to fill in the "Wound Healing Process and Care Information Form" and the "Student Information Form". Then, the wound healing process course will be given as a trainer presentation.
  Interventions: Other: Education
- Experimental 1: The population of the study will consist of students enrolled in the Surgical Diseases Nursing course in the fall and springs semester of the 2022-2023 academic year in the Department of Nursing at the Faculty of Health Sciences of Karadeniz Technical University. The students enrolled in the Surgical Diseases Nursing course in the fall semester will form the control group, while the students enrolled in the spring semester will form the experimental group.

INTERVENTIONS:
Other: Education — Education
  Groups: Control grup 1

SUMMARY:
The goal of this randomized controlled study is to evaluation the effect of mobile application-based wound healing course on clinical reasoning skills in nursing student. The main questions it aims to answer are:

* Does microlearning-based courses have an effect on clinical reasoning skills of nursing students compared to traditional courses?
* Does microlearning-based courses have an effect on the retention of knowledge in nursing students compared to traditional courses? Participants will consist of students enrolled in the Surgical Diseases Nursing course in the fall and springs semester of the 2022-2023 academic year in the Department of Nursing at the Faculty of Health Sciences of Karadeniz Technical University.

If there is a comparison group: Researchers will compare experimental group to see if control group.

DETAILED DESCRIPTION:
Today, there is a need to integrate rapidly developing technology into educational environments and to structure educational environments. Micro-learning modules have been used in e-learning platforms recently, with short content and user focus. This randomized controlled study was planned to evaluation the effect of mobile application-based wound healing course on clinical reasoning skills of nursing students. The population of the study will consist of students enrolled in the Surgical Diseases Nursing course in the fall and springs semester of the 2022-2023 academic year in the Department of Nursing at the Faculty of Health Sciences of Karadeniz Technical University. The students enrolled in the Surgical Diseases Nursing course in the fall semester will form the control group, while the students enrolled in the spring semester will form the experimental group. Students in the control group will take the wound healing process course with the presentation of the trainer, and the students in the experimental group will take micro-learning courses. Data will be collected with the "Student Information Form", "Wound Healing Process Information Form" and "Micro-Learning Based Mobile Application Evaluation Form". In addition, students will be evaluated on the simulator of clinical decision-making processes. The micro-learning course will remain open to students in the experimental group for 31 day. In order to measure the permanence of the knowledge, the "Wound Healing Process Information Form" will be filled in again after 31 days to the students in the control and experimental groups in line with the literature. In addition, students will be evaluated on the simulator of clinical decision-making processes. The results obtained after the application will be analyzed and the effect of the micro-learning course on the decision-making processes of the students will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Enrolling in the Surgical Diseases Nursing course for the first time, Being willing to participate in the study, Having Android or IOS system on the mobile phone.

Exclusion Criteria:

* Having preliminary training and experience in wound care and non-healing (health vocational high school graduation, etc.),

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population of the study will consist of students enrolled in the Surgical Diseases Nursing course in the fall and springs semester of the 2022-2023 academic year in the Department of Nursing at the Faculty of Health Sciences of Karadeniz Technical University.
Sampling Method: Probability Sample
Enrollment: 82 (Estimated)
Dates: Start 2022-10-06 (Actual); Primary Completion 2023-10-10 (Estimated); Study Completion 2023-12-10 (Estimated)

PRIMARY OUTCOMES:
Control group 1 | 2022
  Survey 1
Experimental group 1 | 2023
  Survey 1

SECONDARY OUTCOMES:
Control group 2 | 2022
  Survey 2
Experimental group 2 | 2023
  Survey 2

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin GÜNER, Principal Investigator — yaseminguner@ktu.edu.tr
Locations (1):
- Yasemin GÜNER, Ortahisar, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2022-04-10): https://cdn.clinicaltrials.gov/large-docs/35/NCT05942235/Prot_000.pdf